CLINICAL TRIAL: NCT05485272
Title: Clinical Evaluation of Silver Diamine Fluoride Combined With Potassium Iodide Versus Silver Diamine Fluoride in Management of Class I Carious Lesions Over a Period of 12 Months Follow-up: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of SDF Combined With KI Versus SDF in Management of Class I Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shorouk Hisham Helmy, A Master's Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422019469442
Record Dates: First submitted 2022-07-30; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Carious Lesion
MeSH Terms: conditions — Dental Caries | interventions — Potassium Iodide; silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: A 3-arm randomized clinical trial. Randomization will be done according to a check list including the number of participants divided into 3 groups of 14 patients (42 total) according to interventions/Control assessment methods.
Who Masked: Participant, Outcomes Assessor
Masking Description: The operator will not be blinded due to differences between both materials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention 1 (Experimental): Silver Diamine Fluoride combined with Potassium Iodide (Riva Star), under High-Viscosity Glass Ionomer (EQUIA).
  Interventions: Other: Silver Diamine Fluoride combined with Potassium Iodide.
- Intervention 2 (Experimental): Silver Diamine Fluoride (SDF), under High-Viscosity Glass Ionomer (EQUIA).
  Interventions: Other: Silver Diamine Fluoride.
- The comparator (Active Comparator): High-Viscosity Glass Ionomer (EQUIA).
  Interventions: Other: High-Viscosity Glass Ionomer.

INTERVENTIONS:
Other: Silver Diamine Fluoride combined with Potassium Iodide. — Riva Star, Silver diamine fluoride 38% and potassium iodide, SDI, Bayswater, Australia.
  Other Names: Riva Star.
  Arms: Intervention 1
Other: Silver Diamine Fluoride. — A clear liquid that combines the antibacterial effects of silver and the remineralizing effects of fluoride.
  Other Names: SDF.
  Arms: Intervention 2
Other: High-Viscosity Glass Ionomer. — A Glass Hybrid material.
  Other Names: EQUIA
  Arms: The comparator

SUMMARY:
To evaluate the clinical performance of High-Viscosity Glass Ionomer (EQUIA) versus Silver Diamine Fluoride combined with Potassium Iodide (Riva Star) and Sliver Diamine Fluoride (SDF) under High-Viscosity Glass Ionomer (EQUIA) in deep class I carious lesions, over a period of one year follow-up. The null hypothesis tested in this study, that in deep class I carious lesions, the High-Viscosity Glass Ionomer (EQUIA) versus Silver Diamine Fluoride combined with Potassium Iodide (Riva Star) and Sliver Diamine Fluoride (SDF) under High-Viscosity Glass Ionomer (EQUIA) will show the same clinical performance.

DETAILED DESCRIPTION:
A sample of adults with an age range of 18-40 years old, having a permanent molar with deep class I carious lesions, according to the international caries detection and assessment system (ICDAS), occlusal caries that scored 4 (underlying dark shadow from dentin), or 5 (Distinct cavity with visible dentin), will be selected from the patients attending at the Conservative and Esthetic Dentistry Department Clinic, Faculty of Dentistry, Cairo University, and those who meet the study inclusion criteria will be recruited.

All selected 42 permanent molars will be randomly equally allocated into three groups according to the material used. Group I (n=14) Silver Diamine Fluoride combined with Potassium Iodide (Riva Star) under High-Viscosity Glass Ionomer (EQUIA), Group II (n=14) Silver Diamine Fluoride (SDF) both under High-Viscosity Glass Ionomer (EQUIA), and Group III (n=14) High-Viscosity Glass Ionomer (EQUIA).

Steps in Short:

1. Recruitment of the patients and full examination with diagnosis.
2. Informed consent taking for the eligible participants to participate in the study.
3. Randomization and allocation into three groups.
4. Application of the intervention 1; Silver Diamine Fluoride combined with Potassium Iodide (Riva Star). Intervention 2; Silver Diamine Fluoride (SDF). Both under High-Viscosity Glass Ionomer (EQUIA). The comparator; High-Viscosity Glass Ionomer (EQUIA). All materials were manipulated according to the manufacturers' instructions.
5. Baseline data collection of the clinical evaluation of the restorations using FDI criteria.
6. Follow up at 3, 6, and 12 months for data collection of the clinical evaluation of the restorations using FDI criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with deep class I carious lesions in molars, according to the international caries detection and assessment system (ICDAS), occlusal caries that scored 4 (underlying dark shadow from dentin), or 5 (Distinct cavity with visible dentin).
2. Adults males or females.
3. Age: 18-40 years old.
4. Good Oral hygiene.
5. Co-operative patients, approving to participate in the study.
6. Teeth planned to be restored should be vital.
7. Presence of favorable occlusion.

Exclusion Criteria:

1. Patients having severe systemic diseases, allergies, or adverse medical histories.
2. Patients complaining of sever or active periodontal disease.
3. Lack of compliance.
4. Teeth diagnosed with irreversible pulpitis.
5. Non vital teeth.
6. Heavy occlusion.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Biological Properties: (Postoperative hyper-sensitivity) | 12 Months.
  will be ranked according to Federation Dentaire Internationale criteria (FDI). Scoring system (1,2,3,4,5) by patient interviewing

SECONDARY OUTCOMES:
Functional Properties: (Radiographic examination and Patient's view) (Radiographic examination, and Patient's view) | 12 months.
  will be ranked according to Federation Dentaire Internationale criteria (FDI). Scoring system (1,2,3,4,5) by standardized periapical digital radiographs taken by parallel technique and by patient interviewing
Esthetic: Tooth Color | 12 months.
  by Easy Shade. measuring unit: ΔE

CONTACTS AND LOCATIONS:
Overall Officials: Shorouk H Helmy, Principal Investigator — Cairo University
Locations (1):
- Faculty Of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
after 1 year.